CLINICAL TRIAL: NCT03027713
Title: Diaphragmatic Activity During a Postoperative Rapid Weaning Protocol With Neurally Adjusted Ventilatory Assist in Healthy Lung Patients, a Pilot Study.
Brief Title: Diaphragmatic Activity During Weaning With NAVA, a Pilot Study (NAVA: Neurally Adjusted Ventilatory Assist)
Acronym: NAVA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación para la Investigación del Hospital Clínico de Valencia (Other)
Responsible Party: Principal Investigator, F Javier Belda, Prof. Dr., Fundación para la Investigación del Hospital Clínico de Valencia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: dawNAVA
Record Dates: First submitted 2016-09-04; First posted 2017-01-23 (Estimated); Last update posted 2017-01-23 (Estimated); Status verified 2017-01

CONDITIONS: Postoperative Patients
Keywords: NAVA: neurally adjusted ventilatory assist; Diaphragm electromyographic activity; Weaning

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NAVA group with a specific catheter (Other): The patients were allocated in the NAVA weaning protocol group
  Interventions: Procedure: weaning protocol
- PSV group without a specific catheter (Other): The patients were allocated in the PSV (pressure-support ventilation) weaning protocol group
  Interventions: Procedure: weaning protocol

INTERVENTIONS:
Procedure: weaning protocol — The patients were allocated in the NAVA weaning protocol group o in the PSV weaning protocol group

SUMMARY:
The purpose of this study is to describe the diaphragm electromyographic activity (Edi) in healthy lung patients due to obtain a reference to guide the weaning in those patients

DETAILED DESCRIPTION:
We obtained the Edi recording data at each NAVA level during the weaning in NAVA group, and we compared the respiratory parameters between the PSV and NAVA groups

ELIGIBILITY:
Inclusion Criteria:

* Patients who were scheduled for elective major surgery in which admission to the CCU (critical care unit) for postoperative care and short-term mechanical ventilation with rapid weaning were anticipated.

Exclusion Criteria:

* Preoperative altered central nervous system, neuromuscular or lung disease and ASA (american society of anesthesiologists) classification group IV or NYHA (New York heart association) class IV in the case of cardiac patients. At the CCU, before randomisation, we also excluded patients requiring reoperation, and those who exhibited significant postsurgical bleeding, the development of myocardial infarction, and hemodynamic instability.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-06; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Diaphragmatic electromyographic activity description | 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: Mar Garzando Civera, M.D., Ph.D., Principal Investigator — Fundación para la investigación del Hospital Clínico Universitario de Valencia

IPD SHARING:
Plan to Share IPD: Yes
Shared data will be anonymous